CLINICAL TRIAL: NCT01269645
Title: Evaluating Educational Materials About Cancer Clinical Trials
Brief Title: Facts and Attitudes About Clinical Trials
Acronym: FACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-15820
Record Dates: First submitted 2010-12-22; First posted 2011-01-04 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Cancer; Neoplasm
Keywords: Cancer; Clinical trials
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Usual care and provision of National Cancer Institute brochure "Taking Part in Cancer Treatment Research Studies." Participants will be asked to read this brochure after completion of the baseline surveys and will be given a copy to take home with them.
  Interventions: Behavioral: Clinical Trial educational materials
- Clinical Trial educational materials (Experimental): Usual care and (1) a 10-minute clinical trials educational video; and (2) a 12-page educational booklet to accompany the educational video. Content includes basic information about clinical trials and patient testimonials about the value and benefits of participating in clinical trials. The video also addresses common misperceptions about clinical trials using patient and physician testimonials. After watching the video, participants will be provided a copy of the video for home viewing, along with the educational booklet to be reviewed at home.
  Interventions: Behavioral: Clinical Trial educational materials

INTERVENTIONS:
Behavioral: Clinical Trial educational materials — Usual care and (1) a 10-minute clinical trials educational video; and (2) a 12-page educational booklet to accompany the educational video. Content includes basic information about clinical trials and patient testimonials about the value and benefits of participating in clinical trials. The video also addresses common misperceptions about clinical trials using patient and physician testimonials. After watching the video, participants will be provided a copy of the video for home viewing, along with the educational booklet to be reviewed at home.
  Other Names: Clinical Trials: Are They Right for You?

SUMMARY:
The primary objective of this project is to examine the impact of providing cancer patients with audiovisual information about clinical trials on attitudes towards clinical trial participation. It is hypothesized that patients provided these materials will have more favorable attitudes toward clinical trial participation compared to patients not provided these materials.

Participants will be randomized to either: (1) an intervention condition in which they will be asked to view a short video and read an accompanying brochure about clinical trials developed by the investigative team; or (2) a control condition in which they will be asked to read the National Cancer Institute's brochure entitled "Taking Part in Cancer Treatment Research Studies." Self-report data will be collected at two timepoints: 1) in person following study enrollment, but before receipt of material related to intervention assignment (baseline/Time 1), and 2) by telephone interview between 7 and 28 days following study enrollment (follow-up/Time 2). In addition, data will also be collected from medical records six weeks after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with cancer
2. Have not been asked previously to participate in a clinical trial of a treatment for cancer
3. Be scheduled for a visit with a medical oncologist at the time of recruitment

Exclusion Criteria:

1. Are under the age of 18
2. Do not speak and read standard English
3. Are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2009-07; Primary Completion 2011-09 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to follow-up in attitudes towards clinical trial participation | Baseline (before first med onc visit; after first med onc visit; or before second med onc visit) and Follow-up (7-28 days after baseline)
  The primary objective of this project is to examine the impact of providing cancer patients with audiovisual information about clinical trials on attitudes towards clinical trial participation. It is hypothesized that patients provided these materials will have more favorable attitudes toward clinical trial participation compared to patients not provided these materials.

SECONDARY OUTCOMES:
Impact of information on knowledge, self-efficacy, receptivity, and likelihood of participating | Baseline (before first med onc visit; after first med onc visit; or before second med onc visit) and Follow-up (7-28 days after baseline)
  The secondary objectives are to examine the impact of audiovisual information about clinical trials on knowledge, self-efficacy, receptivity, and likelihood of participating in a clinical trial. It is hypothesized that patients provided audiovisual materials will be more knowledgeable about clinical trials, will believe themselves to be more capable of participating in a clinical trial, will be more receptive to learning more about a clinical trial, and will report greater likelihood of participating in a clinical trial if asked compared to patients not provided these materials.
Impact of information on participation in clinical trials | Medical record review (6 weeks after completion of baseline survey)
  The tertiary objective is to explore the impact of providing cancer patients with audiovisual information about clinical trials on actual participation in clinical trials. Since this aim is exploratory, no hypothesis is offered.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Jacobsen, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (7):
- United States (7):
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Gainesville, Florida
  - Center for Cancer Care & Research/Watson, Lakeland, Florida
  - Ocala Oncology Center, Ocala, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Space Coast Medical Associates, Titusville, Florida
  - Billings Clinic, Billings, Montana